CLINICAL TRIAL: NCT00649064
Title: A Multi-Center Study To Examine The Clinical Effects Of Cross Titration Of Antipsychotics With Ziprasidone In Subjects With Schizophrenia Or Schizoaffective Disorder
Brief Title: A Study of the Effects of Ziprasidone for the Treatment of Schizophrenia or Schizoaffective Disorder in Patients Who Were Switched From Other Antipsychotic Drugs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281120
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizoaffective Disorder; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ziprasidone (Experimental)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — Ziprasidone 40 mg capsules twice daily for the first 7 days followed by flexible dosing between 40 and 80 mg twice daily for the remaining 5 weeks.
  Other Names: Geodon, Zeldox

SUMMARY:
The purpose of this study is to see if differences exist in outcome in patients with schizophrenia or schizoaffective disorder who were switched from other antipsychotics to ziprasidone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Outpatients for at least 3 months on treatment with sulpiride, olanzapine, quetiapine, or risperidone and at least a partial beneficial response to typical antipsychotic treatment including for the current episode
* Partial improvement in symptoms that justified a switch to ziprasidone

Exclusion Criteria:

* Diagnosis of major depression or occurrence of moderate depressive symptoms
* Resistance to conventional antipsychotic drugs
* Treatment with other drugs such as antiseizure medications, antipsychotics, antidepressants, or mood stabilizing agents that might interfere with the assessement of the efficacy of ziprasidone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-12; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Brief Psychiatric Rating Scale (BPRS) total score | Week 6

SECONDARY OUTCOMES:
Adverse events | Weeks 1, 2, and 6
Change from baseline in weight | Baseline and Week 6
Change from baseline in prolactin and lipid levels | Baseline and Week 6
Change from baseline in electrocardiogram | Baseline and Week 6
Change from baseline in Positive and Negative Symptom Scale (PANSS), including PANSS total scores and PANSS positive, PANSS negative, and PANSS general subscale scores | Baseline and Weeks 1, 2, and 6
Change from baseline in Clinical Global Impressions-Severity (CGI-S) scale scores | Baseline and Weeks 1, 2, and 6
Clinical Global Impressions-Improvement (CGI-I) scale scores | Baseline (using historical data) and Weeks 1, 2, and 6
Change from baseline in movement disorder rating scales, including Barnes Akathisia Scale (BAS) and Abnormal Involuntary Movement Scale (AIMS) | Baseline and Week 6
Change from baseline in vital signs | Baseline and Weeks 1, 2, and 6
Change from baseline in Montgomery Asberg Depression Rating Scale (MADRS) scores | Baseline and Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Taiwan (3):
  - Pfizer Investigational Site, Changhua
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281120&StudyName=A%20study%20of%20the%20effects%20of%20ziprasidone%20for%20the%20treatment%20of%20schizophrenia%20or%20schizoaffective%20disorder%20in%20patients%20who%20were%20switched%20fro